CLINICAL TRIAL: NCT06799858
Title: Localization of Breast Cancer with the Sirius Pintuition Magnetic Seed: a Pilot Study in the Czech Republic
Brief Title: Localization of Breast Cancer with the Sirius Pintuition Magnetic Seed
Status: Recruiting | Type: Observational
Sponsor: Jan Žatecký (Other)
Responsible Party: Sponsor-Investigator, Jan Žatecký, Jan Žatecký, MD, PhD, Principal Investigator, Silesian Hospital in Opava
Organization: Silesian Hospital in Opava (Other)
Other Study IDs: EK SNO 429/2024
Record Dates: First submitted 2025-01-22; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Device: Breast cancer localisation with magnetic seed Sirius Pintuition — Patients with histologically proven non-palpable breast cancer or with histologically proven pathological lymph node will be localised by a magnetic seed Sirius Pintuition.

SUMMARY:
A prospective pilot study in the Czech Republic examining the use of magnetic seed Sirius Pintuition for the localization of non-palpable malignant breast tumors and pathological lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer confirmed by a core-cut biopsy
* localisation of non-palpable breast cancer or pathological lymph node with a magnetic seed Sirius Pintuition
* breast cancer surgery in Surgical dpt, Silesian Hospital in Opava

Exclusion Criteria:

* disagree with participation in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-palpable breast cancer or pathological lymph node localised by magnetic seed Sirius Pintuition.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Hypotesis 1 | 1 year
  Localization of non-palpable breast tumors and pathological lymph nodes with a magnetic seed Sirius Pintuition is comparable to other localization methods (iodine seed, wire-guided localisation) in the incidence of complications during intraoperative marker detection (absolute and relative incidence; %).
Hypotesis 1_1 | 1 year
  Localization of non-palpable breast tumors and pathological lymph nodes with a magnetic seed Sirius Pintuition is comparable to other localization methods (iodine seed, wire-guided localisation) in the incidence of complications during marker insertion (absolute and relative incidence; %).
Hypotesis 1_2 | 1 year
  Localization of non-palpable breast tumors and pathological lymph nodes with a magnetic seed Sirius Pintuition is comparable to other localization methods (iodine seed, wire-guided localisation) in the incidence seed migration (absolute and relative incidence, %).

SECONDARY OUTCOMES:
Hypotesis 2 | 1 year
  Localization of non-palpable breast tumors with a magnetic seed Sirius Pintuition is more accurate in terms of more frequent achievement of R0 resection while preserving the oncological radicality (absolute and relative incidence; %).
Hypotesis 2_1 | 1 year
  Localization of non-palpable breast tumors with a magnetic seed Sirius Pintuition is more accurate in removing smaller tissue volume while preserving the oncological radicality (volume, cm3).

CONTACTS AND LOCATIONS:
Locations (1):
- Silesian Hospital in Opava, Opava, Czechia